CLINICAL TRIAL: NCT01053286
Title: Stimulation of Sensation and Improvement in Swallowing Using Oral Capsaicin
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200917225
Record Dates: First submitted 2009-10-20; First posted 2010-01-21 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia; Gastroesophageal Reflux
Keywords: Dysphagia; Globus; Gastroesophageal reflux
MeSH Terms: conditions — Deglutition Disorders; Gastroesophageal Reflux; Globus Sensation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a research study to learn more about whether capsaicin, a natural ingredient of chili peppers that makes them taste "hot", can improve swallowing function. The purpose of this study is to evaluate whether sucking on a capsaicin lozenge improves sensation in the throat enough to improve swallowing function.

DETAILED DESCRIPTION:
Swallowing problems are encountered frequently in primary practice and in the hospital setting. The list of possible causes is large, ranging from strokes and neurological disease through to complications of cancer treatment, acid reflux, and surgery. Many patients have a reduced ability to feel food and fluid (reduced sensation) within the throat (pharynx) and this leads to inability to manipulate food and fluids in the correct manner. This can produce a variety of swallowing problems such as choking on foods and fluids, regurgitation, aspiration, weight loss, malnutrition and poor quality of life.

Treatment is largely directed at rehabilitation of muscle power and education about safe swallowing techniques or positioning that limits food and fluid entering the airway. A novel approach is to try to improve sensation within the pharynx so that patients can feel substances present and then manipulate them in a more appropriate and safe manner. In this regard capsaicin, a nutritional supplement derived from peppers, has shown a stimulatory effect on sensory nerves and an ability to improve the swallowing reflex (Ebihara et al., 2005). Although studies have shown that capsaicin can improve the swallowing reflex, data regarding improvement in swallowing function is lacking. Using a small dose of capsaicin administered as a lozenge, we hope to stimulate sensation within the pharynx enough to improve physical swallowing measures on a contrast swallow study. This method of application is comfortable, easy and directed to the site of action.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Patients with the following condition: dysphagia, globus, gastroesophageal reflux, neurological disease affecting swallowing or any other condition requiring dynamic swallow study
* Patients willing to provide written informed consent for their participation in the study

Exclusion Criteria:

* Patients unable to complete a full dynamic swallow study protocol
* Patients enrolled in another investigational clinical trial that interferes with any testing or testing results
* Patients who are pregnant
* Patients with known sensitivities or allergies to capsaicin or peppers, or nightshades (tomato, bell pepper, eggplant) or latex
* Patients who are prisoners
* Patients who are unable to keep a capsaicin lozenge in their mouth safely for 5 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Otolaryngology clinic
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improvement in sensation and swallowing after using oral capsaicin | Outcome measure will be determined during the conduction of the dynamic swallow study
  Pt will undergo a standard protocol for conducting dynamic swallow studies with the use of increasing increments of liquid barium, followed by paste consistency and solid consistency barium items, then large volume and continuous drinking of barium. Pictures are taken in both lateral and anteroposterior views. Patients enrolled in the study will undergo the usual protocol but instead of the straw drinking large volume liquid bolus, they will first receive the capsaicin 0.1mg lozenge then after sucking that for 5 minutes will swallow a second 20cc bolus of liquid contrast agent in lateral view. The lozenge is an FDA approved food nutritional supplement and is available in several forms over-the-counter without a prescription. The capsaicin lozenge we will use will be a 0.1mg lozenge. This is a very small concentration of the supplement. We expect this to take no more than 5 minutes to fully dissolve. They will then finish the protocol (AP views) as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Belafsky, MD, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States